CLINICAL TRIAL: NCT05038488
Title: A Phase 2a Randomized Controlled Trial of MIB-626 (NAD-boosting Drug) vs. Placebo in Adults With COVID-19 Infection and Early Acute Kidney Injury
Brief Title: Phase 2a MIB-626 vs. Placebo COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Metro International Biotech, LLC (Industry)
Responsible Party: Principal Investigator, Shalender Bhasin, Principal Investigator, Metro International Biotech, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIB-626-202
Record Dates: First submitted 2021-03-18; First posted 2021-09-09 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Covid19; Stage 1 Acute Kidney Injury
Keywords: MIB-626; Covid19; Early Acute Kidney Injury; NAD-boosting drug
MeSH Terms: conditions — COVID-19; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: This will be a two center, randomized, double-blind, placebo- controlled, parallel group, efficacy trial to determine the efficacy of MIB-626 treatment relative to placebo in adult patients with COVID-19 infection and stage 1 acute kidney injury. Participants will be screened for eligibility and those meeting eligibility criteria will be offered participation in the study. The subjects will be randomized by minimization to receive MIB-626 or placebo twice daily for up to 14 days. The participants will be followed for 28 days after the administration of the last dose of the investigational product. Kidney function will be ascertained by daily measurements of serum creatinine, which is the standard of care in hospitalized patients with COVID-19.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MIB-626 (Experimental): Oral administration of MIB-626 substantially raises the intracellular NAD+ levels and activates signaling mechanisms that regulate inflammation and cell survival, downregulates the NLRP3 inflammasome, and attenuates the inflammatory response in a number of experimental models, and protects against tissue damage induced by pro-inflammatory cytokines.
  Interventions: Drug: MIB-626
- Placebo Tablet (Placebo Comparator): A placebo control will be supplied. Participants randomized to placebo will receive matching tablet.
  Matching placebo tablets will be provided by the study's Sponsor, Metro International Biotech, LLC.
  Interventions: Drug: Placebo
- Home Treatment (Other): Participants, who are discharged from the hospital before the completion of the 14-day intervention period, will be provided sufficient study medication to take home with them so they can continue to take the medication twice daily for the remaining duration of the 14-day intervention period.
  Interventions: Drug: MIB-626; Drug: Placebo; Other: Home Treatment

INTERVENTIONS:
Drug: MIB-626 — Fifty participants will be randomized, stratified by sex, remdesivir use, and trial site, in a 3:2 ratio to receive either MIB-626 1.0 g orally or matching placebo twice daily for 14 days.
  Other Names: NAD-boosting drug
  Arms: Home Treatment; MIB-626
Drug: Placebo — Subjects will be randomized to receive either the placebo or 1000-mg MIB-626 twice daily orally.
  Arms: Home Treatment; Placebo Tablet
Other: Home Treatment — Participants, who are discharged from the hospital before the completion of the 14-day intervention period, will be provided sufficient study medication to take home with them so they can continue to take the medication twice daily for the remaining duration of the 14-day intervention period.
  Arms: Home Treatment

SUMMARY:
The proposed phase 2a trial will determine whether MIB-626 treatment in adults with COVID-19 infection and stage 1 acute kidney injury is more efficacious than placebo in preventing worsening of kidney function, as assessed by longitudinal changes in serum creatinine concentration, and in attenuating the inflammatory response to the infection.

DETAILED DESCRIPTION:
This is a two-center, randomized, double-blind, placebo-controlled, parallel-group, phase 2a study that will determine the efficacy and safety of MIB-626 treatment relative to placebo in adult patients with COVID-19 infection and stage 1 acute kidney injury.

Hospitalized adult patients with a confirmed or suspected diagnosis of COVID-19 infection will be screened for conformity to inclusion and exclusion criteria and those meeting eligibility criteria on screening will be offered participation in the study. Fifty participants, who meet all the eligibility criteria, and are able and willing to provide informed consent, will be randomized, stratified by sex, remdesivir use, and trial site, in a 3:2 ratio to receive either MIB-626 1.0 g orally or matching placebo twice daily for 14 days. The participants, who are discharged from the hospital before the completion of the 14-day intervention period, will be provided sufficient study medication to take home with them so they can continue to take the medication twice daily for the remaining duration of the 14-day intervention period.

ELIGIBILITY:
Inclusion Criteria:

* A man or a woman, 18 years or older
* Willing and able to provide informed consent, or with a legal representative who can provide informed consent with participant's assent
* Has Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection confirmed by an approved diagnostic test before randomization
* Currently hospitalized
* Documented increase in serum creatinine of 0.3 mg/dL or 50%-99% over baseline (baseline either based on admission serum creatinine or known pre-admission baseline, defined as most recent previous measurement)
* Participant or legal representative has read and signed the Informed Consent Form (ICF) after the nature of the study has been fully explained
* Is willing and able to provide authorization for the use and disclosure of personal health information in accordance with Health Insurance Portability and Accountability Act (HIPAA)
* Patients who are receiving remdesivir as a part of their clinical care or are in clinical trials of remdesivir or other antiviral drugs may be allowed if they meet other eligibility criteria
* Patients, who are participating in observational studies or studies of nonpharmacological interventions, will be allowed to participate
* Not be pregnant and not planning to become pregnant over the next 6 months

Exclusion Criteria:

* In the intensive care unit at the time of screening or prior to randomization
* Requiring mechanical ventilation at the time of screening or prior to randomization
* Has baseline estimated glomerular filtration rate < 30 ml/min/1.73m2
* Has a history of kidney transplantation or hemodialysis treatment or receiving or expected to receive hemodialysis or peritoneal dialysis at screening and prior to randomization
* Is on mechanical ventilation
* Has a contraindication for MIB-626 or its inert ingredients
* Has a diagnosis of lupus nephritis, polycystic kidney disease, other glomerular disease (other than diabetes)
* Has AST or ALT > 3 times the upper limit of normal
* Has other medical condition which, in the opinion of the Principal Investigator, would jeopardize the safety of the study subject or impact the validity of the study results
* Will exclude patients, who are receiving or are enrolled in placebo-controlled intervention trials of anti-inflammatory or immunomodulatory agents, such as tocilizumab. Occasional use of acetaminophen and nonsteroidal anti-inflammatory drugs, such as ibuprofen, for fever or headache is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum cystatin C levels | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Change from baseline in serum cystatin C levels

SECONDARY OUTCOMES:
Change from baseline to peak concentrations of inflammatory biomarkers (IL6, TNF-alpha, hsCRP, Angiotensin 2 to Angiotensin1, 7 ratio, ACE 2) | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Change from baseline to peak concentrations of inflammatory biomarkers (IL6, TNF-alpha, hsCRP, Angiotensin 2 to Angiotensin1, 7 ratio, ACE 2)
The trajectory of change from baseline in concentrations of inflammatory biomarkers (IL6, TNF-alpha, hsCRP, Angiotensin 2 to Angiotensin1, 7 ratio, ACE 2) | enrollment to 14 days or hospital discharge, or death, whichever comes first
  The trajectory of change from baseline in concentrations of inflammatory biomarkers (IL6, TNF-alpha, hsCRP, Angiotensin 2 to Angiotensin1, 7 ratio, ACE 2)
Change from baseline in markers of endothelial damage (vWF, VCAM, PAI-1) | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Change from baseline in markers of endothelial damage (vWF, VCAM, PAI-1)
Change from baseline in markers of microvascular thrombosis (D-dimer, fibrinogen) | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Change from baseline in markers of microvascular thrombosis (D-dimer, fibrinogen)
The trajectory of change in plasma (NGAL, KIM-1) and urinary (KIM-1, NGAL, albumin) biomarkers of acute kidney injury | enrollment to 14 days or hospital discharge, or death, whichever comes first
  The trajectory of change in plasma (NGAL, KIM-1) and urinary (KIM-1, NGAL, albumin) biomarkers of acute kidney injury
Change in urinary albumin concentration (normalized to urine creatinine) from enrollment to peak during hospitalization | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Change in urinary albumin concentration (normalized to urine creatinine) from enrollment to peak during hospitalization
Change from baseline in oxygen saturation | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Change from baseline in oxygen saturation
Change in high sensitivity troponin-1 concentration from enrollment to peak during hospitalization (measured daily in stored biospecimens) | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Change in high sensitivity troponin-1 concentration from enrollment to peak during hospitalization (measured daily in stored biospecimens)
Change from baseline in intracellular NAD+ concentrations in blood during the 14-day treatment period in a subset of study participants | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Change from baseline in intracellular NAD+ concentrations in blood during the 14-day treatment period in a subset of study participants
Circulating concentrations of MIB-626 and its key metabolites P2Y, NAAD, NAM, 1-methylnicotinamide during the 14-day treatment period | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Circulating concentrations of MIB-626 and its key metabolites P2Y, NAAD, NAM, 1-methylnicotinamide during the 14-day treatment period

OTHER OUTCOMES:
Progression in the stage of acute kidney injury increase in serum creatinine OR serum creatinine > 4.0 mg/dL OR need | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Progression in the stage of acute kidney injury
The WHO 8-point Ordinal Scale of Clinical Status | enrollment to 14 days or hospital discharge, or death, whichever comes first
  The WHO 8-point Ordinal Scale of Clinical Status
Change from baseline in Modified Sequential Organ Failure Assessment (SOFA) Score (SOFA) Score | enrollment to 14 days or hospital discharge, or death, whichever comes first
  Change from baseline in Modified Sequential Organ Failure Assessment (SOFA) Score
The number and proportion of patients requiring mechanical ventilation, hemodialysis, or transferred to ICU | enrollment to 14 days or hospital discharge, or death, whichever comes first
  The number and proportion of patients requiring mechanical ventilation, hemodialysis, or transferred to ICU
The number and proportion of patients requiring hemodialysis | enrollment to 14 days or hospital discharge, or death, whichever comes first
  The number and proportion of patients requiring hemodialysis
The number and proportion of patients who die | enrollment to 14 days or hospital discharge, or death, whichever comes first
  The number and proportion of patients who die
The number of days it takes for the temperature to return to normal (<99F) | enrollment to 14 days or hospital discharge, or death, whichever comes first
  The number of days it takes for the temperature to return to normal (<99F)
The length of hospital stay | enrollment to 14 days or hospital discharge, or death, whichever comes first
  The length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- The Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared

REFERENCES:
- [Derived] Pencina KM, Leaf DE, Valderrabano RJ, Waikar SS, Mehta TS, Shang YV, Latham NK, John T, Volpi E, Fusco D, Memish-Beleva Y, Krishnamurthy S, Lavu S, Karmi S, Livingston DJ, Bhasin S. Oral MIB-626 (beta Nicotinamide Mononucleotide) Safely Raises Blood Nicotinamide Adenine Dinucleotide Levels in Hospitalized Patients With COVID-19 and Acute Kidney Injury: A Randomized Controlled Trial. FASEB Bioadv. 2025 Jun 18;7(8):e70011. doi: 10.1096/fba.2025-00014. eCollection 2025 Aug. PMID 40746868